CLINICAL TRIAL: NCT04922034
Title: Study of Patient's Outcomes After a Negative Reintroduction Test for Amoxicillin
Brief Title: Outcome of Patients After a Negative Oral Challenge to Amoxicillin
Acronym: REINAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC21_0178
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2021-06

CONDITIONS: Negative Challenge to Amoxicillin
Keywords: penicillins; reintroduction
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Amoxicillin — Outcome of patients with negative oral challenge to amoxicillin

SUMMARY:
This study aims to evaluate the outcome of patients who had a negative oral challenge to Amoxicillin

DETAILED DESCRIPTION:
This is a prospective, single-center, non-interventional study of patients with negative Amoxicillin oral challenge performed at Angers University Hospital between 2017 and 2019.

An information letter indicating the purpose of the study is sent to eligible patients. If they do not object, patients are contacted by telephone to answer the questionnaire. This questionnaire concerns the reintroduction of penicillins at home after the challenge.

ELIGIBILITY:
Inclusion Criteria:

* Patients whith a negative challenge to Amoxicillin in the Allergology Department of the CHU of Angers between 2017 and 2019.
* Major patients.

Exclusion Criteria:

* Poor comprehension of the French language or cognitive disorders affecting the reliability of the questionnaire
* Person objecting to participate in this research and to the processing of their medical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, single-center, non-interventionnel study of patients with a negative oral challenge to Amoxicillin at Angers University Hospital between 2017 and 2019.
  An information letter indicating the purpose of the study is sent to eligible patients. If they do not object, patients are contacted by telephone one month after the information letter is sent, to answer the questionnaire. This questionnaire, filled in during the telephone interview, concerns the resumption or not of penicillins since the reintroduction test.
  This study concerns all patients, agreeing to participate in this study, who had a negative challenge test to Amoxicillin at the CHU of Angers from 2017 to 2019.
  The potential inclusion is approximately 200 individuals.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Resumption of Amoxicillin after a negative oral challenge to Amoxicillin | Oral challenge test oxxuring between 2017 and 2019, and follow-up until the day of the call
  The main objective is to know if patients who had a negative test for reintroduction of Amoxicillin, have resumed this molecule afterwards.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Angers, Maine Et Loire, France